CLINICAL TRIAL: NCT07158034
Title: Investigating EEG as a Biomarker for Tinnitus Improvement After Bimodal Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025649
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Use Lenire device for 1 hour daily
  Interventions: Device: Lenire Device
- Control Group (No Intervention): Participants in the control group will not receive the stimulation device and will not undergo any stimulation during the study.

INTERVENTIONS:
Device: Lenire Device — The Lenire device is a non-invasive stimulation system designed to reduce the symptoms of chronic subjective tinnitus. It includes a controller that is connected to headphones for sound delivery to the ears and a mouthpiece that provides mild electrical stimulation to the surface of the tongue. Users are recommended to use the device for 60 minutes daily, either in two consecutive 30-minute sessions or at different times throughout the day, for a minimum of 36 hours.
  Arms: Treatment Group

SUMMARY:
The aim of the proposed study is to investigate the use of resting-state Electroencephalogram (EEG)-Based Brain Entropy (EBDBE) and auditory brainstem responses (ABR) as an objective measure of tinnitus improvement following the use of a bimodal stimulation device in individuals with tinnitus after six weeks of bi-modal stimulation.

ELIGIBILITY:
Treatment Group Inclusion Criteria:

* 18 years and over at time of consent
* Ability to read and understand English
* Willing and able to provide and understand informed consent
* Willing to commit to the full duration of the investigation
* Subjective tinnitus
* Tinnitus duration of greater than or equal to 3 months and less than or equal to 20 years at time of consent (only for participants in treatment group)
* Baseline THI score from 40 to 76 (only for participants in treatment group)
* Hearing loss condition - can hear the acoustic stimulation of the Lenire device (only for participants in treatment group)

Treatment Group Exclusion Criteria:

* Subjective tinnitus, where pulsatility is the dominant feature (only for participants in treatment group)
* Objective tinnitus
* Can't hear acoustic stimulation of the Lenire device within its mid- range volume setting
* Began wearing hearing aids within the past 3 months
* A healthcare provider has diagnosed Meniere's disease or another disorder associated with fluctuating hearing loss.
* History of auditory hallucinations
* Tumor on the hearing or balance nervous systems
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* Initiated new prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Ceased prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Changed dosage of prescription medications in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Any use of benzodiazepines or sedative hypnotics (either regularly or on demand)
* Neurological condition that may lead to seizures or loss of consciousness (e.g., epilepsy)
* Participant with a pacemaker or other electro-active implanted device
* Participant previously diagnosed with psychosis or schizophrenia
* Participants diagnosed with Burning Mouth Syndrome
* A diagnosis of bothersome temporomandibular joint disorder (TMJ) has been rendered
* Previous involvement in a clinical investigation for tinnitus treatment or had an implantable or surgical intervention for tinnitus
* Inability to physically or comprehensively use the device
* Oral piercings that cannot or will not be removed
* Pregnancy per patient report
* Prisoner
* PI does not deem the candidate to be suitable for the investigation for other reasons not listed above. Rationale must be provided.

Control Group Inclusion Criteria:

* 18 years and over at time of consent
* Ability to read and understand English
* Willing and able to provide and understand informed consent
* Willing to commit to the full duration of the investigation

Control Group Exclusion Criteria:

* Began wearing hearing aids within the past 3 months
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* Initiated new prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Ceased prescription medications or medical treatments in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Changed dosage of prescription medications in the previous 3 months that may impact the outcomes of the investigation, based on class of medication: antidepressants, anticonvulsants, neuroleptics and opioid analgesics.
* Any use of benzodiazepines or sedative hypnotics (either regularly or on demand)
* Neurological condition that may lead to seizures or loss of consciousness (e.g., epilepsy)
* Participant previously diagnosed with psychosis or schizophrenia
* A diagnosis of bothersome temporomandibular joint disorder (TMJ) has been rendered
* Prisoner
* PI does not deem the candidate to be suitable for the investigation for other reasons not listed above. Rationale must be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in brain waves at 6 weeks | Week 6
  Assessed via 32-channel EEG recording

SECONDARY OUTCOMES:
Correlation between change in EBDBE, ABR, THI, and PSS-10 | Week 6
  Assessed via Tinnitus Handicap Inventory (THI) and Perceived Stress Scale (PSS), for which lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Nelson, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No